CLINICAL TRIAL: NCT05007691
Title: Single-group, Comparative Biomechanical Study of Maxillary and Mandibular Splints Used for the Treatment of Masticatory Muscle Parafunction
Brief Title: Comparative Study of Maxillary and Mandibular Splints Used for the Treatment of Masticatory Muscle Parafunction (FEA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Arutyunov-2
Record Dates: First submitted 2021-08-10; First posted 2021-08-16 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2021-07

CONDITIONS: Jaw, Edentulous; Mouth, Edentulous
Keywords: Denture, Complete; Technology, Dental; Biomedical and Dental Materials
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: patients are included in a single study group. In a study group, each patient is assessed for both of the same primary treatment. The final results for each of the treatments for each patient are used for further analysis by the finite element method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Occlusal splints (Experimental): In a clinical setting, participants test the closure of the occlusal splint with the antagonistic dentition.
  Only one of the two occlusal splints (mandibular splint and maxillary splint) is used at a time. Occlusal splints are applied separately and alternately.
  Interventions: Device: Occlusal splint

INTERVENTIONS:
Device: Occlusal splint — Occlusal splints are hard, made of polymer biocompatible material using digital additive technology.

SUMMARY:
the purpose of this study is to clarify the rationale for the choice of the upper or lower jaw for positioning the occlusal splint

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients are giving written informed consent. Occlusal splints for the upper and lower jaws are made for each of the patients. An assessment is made of the relative values and distribution of chewing forces in two cases:

1. "maxillary occlusal splint - lower dentition";
2. "mandibular occlusal splint - upper dentition". The obtained values are used in the final elemental analysis of the stress-strain state and the degree of displacement of the dentition in both indicated cases.

ELIGIBILITY:
Inclusion Criteria:

* continuous dentition
* diagnosis (by ICD*-10): K03.0 Excessive attrition of teeth
* diagnosis (by ICD-10): K07.6 Temporomandibular joint disorders
* complaints of nocturnal bruxism
* complaints of discomfort in the area of the chewing muscles
* no history of orthopedic and / or orthodontic treatment
* absence of concomitant general somatic pathologies in the stage of decompensation
* no history of psychogenic and psychosomatic disorders
* no history of cancer *ICD - Classification of Diseases

Exclusion Criteria:

* refusal of the patient during the clinical trial from further treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Difference between mandible and maxilla of occlusal splints in terms of stress-strain state and magnitude of displacement of the splinted teeth | during one appointment, up to 2 hours
  By means of the final elemental analysis, data on the stress-strain state (in MPa) and the displacement of the splinted teeth (in mm) will be obtained, individually for each patient.

SECONDARY OUTCOMES:
Difference between mandible and maxilla dentition in terms of stress-strain state and magnitude of displacement of the teeth | during one appointment, up to 2 hours
  By means of the final elemental analysis, data on the stress-strain state (in MPa) and the displacement of the teeth (in mm) will be obtained, individually for each patient.

OTHER OUTCOMES:
Measurement of the influence of the occlusal splint use on the indicators of the stress-strain state and the magnitude of tooth displacement | during one appointment, up to 2 hours
  By means of the final elemental analysis, data on the stress-strain state (in MPa) and the displacement of the teeth (in mm) will be obtained, individually for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Arutyunov, PhD, Study Director — A.I. Yevdokimov Moscow State University of Medicine and Dentistry
Locations (1):
- A.I. Yevdokimov Moscow State University of Medicine and Dentistry, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in temporomandibular joint disorders.
  Data or samples shared will be coded, with no protected health information included.
  Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
  Request will be evaluated under common conditions by Interuniversity Ethics Committee (A.I. Evdokimov Moscow State University of Medicine and Dentistry)
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 6 months after article publication.
Access Criteria: Access to trial IPD (individual participant data) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Gribov D, Antonik M, Butkov D, Stepanov A, Antonik P, Kharakh Y, Pivovarov A, Arutyunov S. Personalized Biomechanical Analysis of the Mandible Teeth Behavior in the Treatment of Masticatory Muscles Parafunction. J Funct Biomater. 2021 Apr 9;12(2):23. doi: 10.3390/jfb12020023. PMID 33918647